CLINICAL TRIAL: NCT04425343
Title: Microbial Profiling in Pockets Related to Chronic Periodontitis Patients in UAE Population Using 16s RNA Metagenomics Sequencing
Brief Title: Microbial Profiling in Pockets Related to Chronic Periodontitis Patients Using 16s RNA Metagenomics Sequencing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajman University (Other)
Responsible Party: Principal Investigator, sudhir rama varma, Assistant Professor, Ajman University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: F-H-17-11-03
Record Dates: First submitted 2020-06-07; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Periodontal Diseases
Keywords: metagenomics; 16S; Periodontitis, Adult
MeSH Terms: conditions — Periodontal Diseases; Chronic Periodontitis

STUDY DESIGN:
Intervention Model Description: . Patients recruited for the study were diagnosed as Stage II Generalized periodontitis according to the classification from the 2017 world workshop on the "classification of periodontal and peri-implant disease and conditions". Periodontal status indicating the severity of interdental clinical attachment loss of 3-4mm, radiographic bone loss between 15%-33% and with no tooth loss were included. The complexity of periodontitis with a maximum probing depth of ≤ 5mm with horizontal bone loss and having an extent and distribution with >30% teeth involved were included in the study.
Who Masked: Investigator
Masking Description: . A total of 80 plaque samples were collected with the clinical characteristics of the patient comprising of age between 25-39 years, 36 females and 44 males
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periodontitis, Adult (Experimental): Plaque samples were taken from subgingival pocket and send to the lab for metagenomic analysis
  Interventions: Genetic: 16s RNA Metagenomics sequencing
- Metgenomic analysis (Experimental): Analysis for whole bacterial count
  Interventions: Genetic: 16s RNA Metagenomics sequencing

INTERVENTIONS:
Genetic: 16s RNA Metagenomics sequencing — The subgingival plaque was collected using a sterile curette from the buccal aspect of maxillary molars and lingual aspect of mandibular incisors, in a vial containing 200µl of Buffer CL.
  Other Names: DNA isolation

SUMMARY:
The study was developed in compliance with the Helsinki Declaration on medical research involving the Ethics Committee at Ajman University (2017-A-DN-04). Informed consent from all the participants was obtained before participation in the study. The participants were systemically healthy with no history of antibiotics for the past three months. Patients recruited for the study were diagnosed as Stage II Generalized periodontitis according to the classification from the 2017 world workshop on the "classification of periodontal and peri-implant disease and conditions". Periodontal status indicating the severity of interdental clinical attachment loss of 3-4mm, radiographic bone loss between 15%-33% and with no tooth loss were included. The complexity of periodontitis with a maximum probing depth of ≤ 5mm with horizontal bone loss and having an extent and distribution with >30% teeth involved were included in the study. A total of 80 plaque samples were collected with the clinical characteristics of the patient comprising of age between 25-39 years, 36 females and 44 males. The subgingival plaque was collected using a sterile curette from the buccal aspect of maxillary molars and lingual aspect of mandibular incisors, in a vial containing 200µl of Buffer CL.

DETAILED DESCRIPTION:
The collected plaque samples were then freshly prepared for the DNA isolation using ABIOpure TM Total DNA (version 2.0) (Cat No: M501DP100) according to the manufacturer's instruction. All the samples were assessed for DNA quantification using spectrophotometry and further quantified using the fluorometric method. This was performed using DeNovix DS-11 FX (DeNovix). Further to the DNA quantification, assessment of DNA integrity was resolved on a 0.8% agarose gel with ethidium bromide. For NGS library preparation, all the samples underwent PCR amplification of the 16S rRNA gene in the isolated bacterial DNA. The primers used had targeted in the V3-V4 region of the 16S rRNA gene. The full length primer sequences, using standard IUPAC nucleotide nomenclature, to follow the protocol targeting this region are:

16SAmpliconPCRForwardPrimer=5' TCGTCGGCAGCGTCAGATGTGTATAAGAGACAGCCTACGGGNGGCWGCAG 16SAmpliconPCRReversePrimer=5' GTCTCGTGGGCTCGGAGATGTGTATAAGAGACAGGACTACHVGGGTATCTAATCC Gel electrophoresis method was used for the size selection and the bioinformatics pipeline used for processing microbiome 16S sequence data was QIIME

ELIGIBILITY:
Inclusion Criteria:

* Patients recruited for the study were diagnosed as Stage II Generalized periodontitis
* Medically fit

Exclusion Criteria:

* Patients having gingivitis or stage III periodontitis
* Medically unfit

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2019-10-07 (Actual)

PRIMARY OUTCOMES:
Microbial Taxonomical Composition | From Baseline to 3 months
  The composition was determined using subgingival plaque samples and performing 16s metagenomic sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Sudhir Varma, MDS, Principal Investigator — Assistant Professor
Locations (1):
- Ajman University of Science and Technology, Ajman, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No
Microbial Taxonomical Composition